CLINICAL TRIAL: NCT06854081
Title: A Multi-Center Registry Evaluating EluPro Antibiotic-Eluting BioEnvelope During CIED Implantation
Brief Title: EluPro Antibiotic-Eluting BioEnvelope Registry
Status: Recruiting | Type: Observational
Sponsor: Elutia Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CPR-2404
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Arrhythmias
Keywords: EluPro; CIED; Envelope; Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- EluPro: EluPro Antibiotic-Eluting BioEnvelope
  Interventions: Combination Product: EluPro Antibiotic-Eluting BioEnvelope

INTERVENTIONS:
Combination Product: EluPro Antibiotic-Eluting BioEnvelope — Utilization of an EluPro Antibiotic-Eluting BioEnvelope with the CIED during the participant's CIED implant procedure.

SUMMARY:
A Multi-Center Registry Study Evaluating Participants Who Receive EluPro Antibiotic-Eluting BioEnvelope During CIED Implantation

DETAILED DESCRIPTION:
This prospective, multi-center registry study will enroll up to 100 participants who will receive an EluPro Antibiotic-Eluting BioEnvelope during their CIED procedure.

Participant data will be captured at several time points: Screening/Enrollment, day of Surgical Procedure, and at Wound Check (2-4 Weeks) 3, 6, and 12 months post-surgery, as well as any unscheduled visits up to 12 months post-surgery. Any follow-up visit can be completed via telephone/video if the participant is not scheduled to be seen in the office. Patient-reported outcomes such as implant site pain and satisfaction questionnaires shall be administered to participants at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing implantation of EluPro with either a de novo CIED implantation or has an existing CIED and is undergoing CIED replacement or upgrade.
* Patient is willing to comply with scheduled follow-up and study-related visits.
* Patient is 18 years of age or older at the time of enrollment.
* Patient agrees to provide written informed consent and use of PHI.

Exclusion Criteria:

* Patient has a prior history of CIED infection, other prosthetic device infection, or endovascular infection, including endocarditis, in the past 12 months.
* Patient is exhibiting signs or symptoms consistent with any type of active infection (including but not limited to pneumonia, urinary tract, cellulitis, or bacteremia).
* Patient has Stage 4 or 5 kidney disease (eGFR <30 ml/min).
* Patient requires long-term vascular access for any reason.
* Patient is undergoing implantation of a CIED that does not fit completely into EluPro, preventing closure of the bioenvelope to secure the CIED.
* Patient is currently on chronic immunosuppressive agents or ≥20mg/day of Prednisone or equivalent.
* Patient has known allergy to minocycline or rifampin or their derivatives, or any other known contraindications to the implantation of EluPro.
* Patient is participating in another clinical study that could impact the outcome and documented pre-approval from the study sponsor has not been obtained.
* Female patient who is pregnant, or of childbearing potential and not on a reliable form of birth control. Women of childbearing potential are required to have a negative pregnancy test within 7 days prior to device procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 100 participants who will receive a EluPro Antibiotic-Eluting BioEnvelope during their CIED procedure
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events/Complication Rates | 12 Months
  Determine the rates of adverse events and complications associated with the use of EluPro device envelope in real-world settings.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UC San Diego Health, La Jolla, California
  - Tallahassee Research Institute, Tallahassee, Florida
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No